CLINICAL TRIAL: NCT06152510
Title: Comparative Study of Static Balance Abilities in Children With Autism and Neurotypical Peers
Brief Title: Static Balance in Children With Autism vs. Neurotypical Peers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: CNR-IRIB-PRO-2023-006
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Autism; virtual reality; virtual reality rehabilitation system; postural control
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with autism spectrum condition: Thirty children with autism spectrum condition and with medium-high functioning, aged 4 to 13 years, IQ > 75, in the absence of motor deficits due to another clinical condition.
  Interventions: Other: Virtual Reality Rehabilitation System
- Children with typical development: Thirty children with typical development aged 4 to 13 years, IQ > 75, in the absence of motor deficits due to clinical condition.
  Interventions: Other: Virtual Reality Rehabilitation System

INTERVENTIONS:
Other: Virtual Reality Rehabilitation System — In a single session to evaluate postural control, both children with ASD and typically developing peers will participate in an activity utilizing the Virtual Reality Rehabilitation System (VRRS) in conjunction with a stabilometric balance platform. During the assessment task, participants will stand on the balance platform with their eyes open, focusing on a fixed point displayed on the VRRS screen for a duration of one minute. This process will be repeated three times for each participant. The combined use of VRRS and the stabilometric balance platform aims to provide a comprehensive evaluation of postural control abilities in both groups, allowing for the observation and measurement of potential differences in stability and balance performance between children with ASD and their neurotypical counterparts.

SUMMARY:
The Virtual Reality Rehabilitation System (VRRS) is an innovative and sophisticated technology, aimed to generate immersive and interactive settings intended for therapeutic and evaluative objectives. Through the utilization of virtual reality technology, it constructs diverse scenarios, tasks, and activities in a controlled digital environment, fostering engagement. Primarily crafted for rehabilitation purposes, the VRRS features adaptable programs addressing various therapeutic requirements, encompassing motor skill enhancement, cognitive challenges, and assessments related to balance.Understanding the nuanced motor abilities in children, particularly those with neurodevelopmental conditions like autism, is a critical area of research in pediatric rehabilitation. The significance of this research lies in comprehending the specific balance challenges experienced by children with autism spectrum disorder (ASD), a population often noted for motor coordination and balance difficulties. Because VRRS offers a controlled and engaging environment, this study seeks to provide a detailed analysis of static balance abilities in capabilities in children diagnosed with ASD in comparison to typically developing (TD) children. The study also wants to explore the efficacy of VRRS as an assessment tool for pediatric balance evaluations.The primary objective of this study is to highlight the distinctions in postural control between ASD and TD children, utilizing an objective quantification tool to delineate the differences between the two groups. This will be achieved through a group comparison study involving two distinct cohorts. The first group will comprise 30 school-aged children with ASD, while the second group will consist of 30 TD school-aged children. To evaluate postural control, both groups will participate in an activity utilizing the VRRS in conjunction with a stabilometric balance platform. During the assessment task, participants will stand on the balance platform with their eyes open, focusing on a fixed point displayed on the VRRS screen for a duration of one minute. This process will be repeated three times for each participant. The combined use of VRRS and the stabilometric balance platform aims to provide a comprehensive evaluation of postural control abilities in both groups, allowing for the observation and measurement of potential differences in stability and balance performance between children with ASD and their neurotypical counterparts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism; QI ≥ 75

Exclusion Criteria:

* Motor deficits due to another clinical condition

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Thirty children with Autism Spectrum Disorder (ASD) and 30 typically developing (TD) children will participate in the study. The children with ASD will be recruited and tested at the clinical facilities of the Institute for Biomedical Research and Innovation of the National Research Council of Italy (IRIB-CNR) in Messina. To be included in the study the child needs to have an ASD diagnosis based on the Diagnostic and Statistical Manual, Fifth Edition (DSM-5) criteria from a licensed clinical child neuropsychiatrist but no established intellectual disability diagnosis. The TD children will recruit through advertisements in schools located close to the Institute. Informed consent will obtain from all subjects involved in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Centre of Pressure (COP) displacement | The test needs approximately 3 minutes per child
  The Virtual Reality Rehabilitation system (VRRS; Khymeia, Italy) is an innovative system based on the concept of augmented feedback. It consists of devices for clinical use and a tablet for home-based telerehabilitation, which can be remotely managed. Different peripherals can be connected via USB to the VRRS, including a stabilometric balance platform. It is a force plate (80 ×55 cm) able to detect forces in the z-direction and the Centre of Pressure (COP) displacement in millimeter (mm). The COP displacement is the distance and direction that COP moves from a reference point or position, in the anterior-posterior (AP) and medial-lateral (ML) direction, thanks to the four load cells integrated into the balance platform. Moreover, a dedicated software can be used to calibrate the balance platform which will allow the estimation of static postural data. After each measurement, a report containing a summary of the data can be exported through the dedicated software.
Centre of Pressure (COP) velocity | The test needs approximately 3 minutes per child
  The Virtual Reality Rehabilitation system (VRRS; Khymeia, Italy) is an innovative system based on the concept of augmented feedback. It consists of devices for clinical use and a tablet for home-based telerehabilitation, which can be remotely managed. Different peripherals can be connected via USB to the VRRS, including a stabilometric balance platform. It is a force plate (80 ×55 cm) able to detect Centre of Pressure (COP) velocity in millimeter per second (mm/s), a sensitive measure to detect changes in postural control.
Centre of Pressure (COP) sway area | The test needs approximately 3 minutes per child
  The Virtual Reality Rehabilitation system (VRRS; Khymeia, Italy) is an innovative system based on the concept of augmented feedback. It consists of devices for clinical use and a tablet for home-based telerehabilitation, which can be remotely managed. Different peripherals can be connected via USB to the VRRS, including a stabilometric balance platform. It is a force plate (80 ×55 cm) able to detect the Centre of Pressure (COP) sway area in square millimeter per second (mm2 /s). Sway area is the area enclosed by the COP trajectory per unit time.
Movement Assessment Battery for Children - Second Edition (MABC-2) | The test needs approximately 40 minutes.
  The Movement Assessment Battery for Children - Second Edition (MABC-2) is an assessment test specifically developed for children from 3 to 16 years with motor function impairment. The tasks are divided by age range and organized into three sections: manual dexterity, aiming and catching and balance. Scores are provided in standard scores and percentiles and are interpreted by using a traffic light system: green light (scores above 15 percentile), meaning typical motor performances; yellow light (scores between 5 and 15 percentile), indicating a risk for motor impairment; red light (scores below 5 percentile), identifying a significant motor function impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beani E, Filogna S, Martini G, Barzacchi V, Ferrari A, Guidi E, Menici V, Cioni G, Sgandurra G. Application of Virtual Reality Rehabilitation System for the assessment of postural control while standing in typical children and peers with neurodevelopmental disorders. Gait Posture. 2022 Feb;92:364-370. doi: 10.1016/j.gaitpost.2021.12.008. Epub 2021 Dec 10. PMID 34923256
- [Background] Kaur M, M Srinivasan S, N Bhat A. Comparing motor performance, praxis, coordination, and interpersonal synchrony between children with and without Autism Spectrum Disorder (ASD). Res Dev Disabil. 2018 Jan;72:79-95. doi: 10.1016/j.ridd.2017.10.025. Epub 2017 Nov 6. PMID 29121516
- [Background] Martini G, Beani E, Filogna S, Menici V, Cioni G, Battini R, Sgandurra G. New Technological Approach for the Evaluation of Postural Control Abilities in Children with Developmental Coordination Disorder. Children (Basel). 2022 Jun 26;9(7):957. doi: 10.3390/children9070957. PMID 35883941